CLINICAL TRIAL: NCT05702086
Title: Evaluating the Utility of a Psychoeducational Serious Game (SPARX) in Protecting Inuit Youth From Depression: A Pilot Study
Brief Title: Making SPARX Fly in Nunavut: Pilot Testing an E-intervention for Boosting Resilience Against Youth Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Collaborators: Government of Nunavut (Unknown); Qaujigiartiit Health Research Centre (Unknown)
Responsible Party: Principal Investigator, Yvonne Bohr, Associate Professor, York University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02 004 15N-M
Record Dates: First submitted 2023-01-10; First posted 2023-01-27 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Depressive Symptoms; Emotion Regulation
Keywords: hopelessness; catastrophizing; rumination; resilience
MeSH Terms: conditions — Depression; Emotional Regulation; Rumination Syndrome | interventions — Gene Expression; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Play now" intervention group (Experimental): The sequence of SPARX play differed for the youth depending on whether they were in Group A ("play now" intervention group) or Group B ("play later" waitlist group). Both groups completed the pre-intervention surveys at Time 1, the beginning of the study. Group A youth then began to play SPARX for seven weeks while Group B waited. During their wait time of seven weeks, Group B youth were not required to participate in any SPARX activities or meet with the community facilitator during their wait period, and they were provided with no additional SPARX-related information. After seven weeks (Time 2), Group A youth completed post-intervention surveys, while Group B youth began their engagement with SPARX by first completing an additional set of pre-intervention surveys, immediately followed by seven weeks of SPARX play. Once Group B youth completed their SPARX gameplay (Time 3), they completed post-intervention surveys.
  Interventions: Other: SPARX (Smart, Positive, Active, Realistic, X-Factor thoughts)
- "Play later" waitlist group (Active Comparator): The sequence of SPARX play differed for the youth depending on whether they were in Group A ("play now" intervention group) or Group B ("play later" waitlist group). Both groups completed the pre-intervention surveys at Time 1, the beginning of the study. Group A youth then began to play SPARX for seven weeks while Group B waited. During their wait time of seven weeks, Group B youth were not required to participate in any SPARX activities or meet with the community facilitator during their wait period, and they were provided with no additional SPARX-related information. After seven weeks (Time 2), Group A youth completed post-intervention surveys, while Group B youth began their engagement with SPARX by first completing an additional set of pre-intervention surveys, immediately followed by seven weeks of SPARX play. Once Group B youth completed their SPARX gameplay (Time 3), they completed post-intervention surveys.
  Interventions: Other: SPARX (Smart, Positive, Active, Realistic, X-Factor thoughts)

INTERVENTIONS:
Other: SPARX (Smart, Positive, Active, Realistic, X-Factor thoughts) — SPARX (Smart, Positive, Active, Realistic, X-Factor thoughts) is a psychoeducational serious game (an e-intervention that utilizes gaming for serious purposes) that teaches established cognitive behavioural therapy strategies and techniques across seven levels or modules. The game is designed to address depressive symptoms in youth by helping them cope with negative thoughts and feelings, represented in the game as GNATs-Gloomy Negative Automatic Thoughts. SPARX was originally designed and developed at the University of Auckland with the specific needs of certain underserved groups of youth in mind, including Māori rangatahi, the Indigenous young people of Aotearoa, New Zealand.

SUMMARY:
The goal of this pilot trial was to test SPARX with Inuit youth in Northern Canada. SPARX is an educational video game designed to teach cognitive behavioural therapy strategies and techniques. This "serious game" has previously shown promise in addressing symptoms of depression with Māori youth in New Zealand. Researchers in this study tested SPARX's suitability with Inuit youth in the territory of Nunavut using surveys that youth completed before and after gameplay.

Hypothesis 1: Youth who completed SPARX were expected to experience a decrease in depressive symptoms and risk factors related to depression. Hypothesis 2: Youth who completed the SPARX program were expected to experience an increase in factors related to resilience.

A team of Nunavut-based community mental health staff facilitated youth's participation in this remote pilot trial with 24 youth aged 13-18 across 11 communities in Nunavut. These youth had been identified by community facilitators as showing low mood, depression, and/or significant levels of stress.

ELIGIBILITY:
Inclusion Criteria:

* one or more of the following:

  * low mood
  * negative affect
  * depressive presentations
  * significant levels of stress and:
  * sufficient English language comprehension to use and understand SPARX

Exclusion Criteria:

None

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2014-09-08 (Actual); Primary Completion 2015-04-22 (Actual); Study Completion 2015-04-22 (Actual)

PRIMARY OUTCOMES:
"Centre for Epidemiologic Depression Scale - Revised" | Pre-gameplay (T=0)
  20-item, self-report scale that aims to measure current depressive symptomatology; total scores range 0-60 with higher score representing worse depression
"Centre for Epidemiologic Depression Scale - Revised" | Post-gameplay (T=7 weeks)
  20-item, self-report scale that aims to measure current depressive symptomatology; total scores range 0-60 with higher score representing worse depression
"Hopelessness Scale for Children" | Pre-gameplay (T=0)
  17 true-false items, which describe negative future expectations and negative present attitudes; scores range from 0-17 with higher score representing greater hopelessness for the future
"Hopelessness Scale for Children" | Post-gameplay (T=7 weeks)
  17 true-false items, which describe negative future expectations and negative present attitudes; scores range from 0-17 with higher score representing greater hopelessness for the future
"Cognitive Emotion Regulation Questionnaire - Short" | Pre-gameplay (T=0)
  18-item measure used with adolescents composed of nine coping styles, which are each coded as separate subscales of emotion regulation; items are scored on a Likert scale (1-5) with higher values corresponding to greater use of that cognitive strategy. Some strategies are positive, others negative
"Cognitive Emotion Regulation Questionnaire - Short" | Post-gameplay (T=7 weeks)
  18-item measure used with adolescents composed of nine coping styles, which are each coded as separate subscales of emotion regulation; items are scored on a Likert scale (1-5) with higher values corresponding to greater use of that cognitive strategy. Some strategies are positive, others negative
"Child and Youth Resilience Measure - Short" | Pre-gameplay (T=0)
  12-item self-report measure that includes three dimensions (Individual, Relational, and Contextual) that reflect the major categories of resilience; total scores range from 12-36 (no; sometimes; yes for 12 items at 1, 2, 3, points respectively); higher scores indicate higher resilience
"Child and Youth Resilience Measure - Short" | Post-gameplay (T=7 weeks)
  12-item self-report measure that includes three dimensions (Individual, Relational, and Contextual) that reflect the major categories of resilience; total scores range from 12-36 (no; sometimes; yes for 12 items at 1, 2, 3, points respectively); higher scores indicate higher resilience

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Bohr, PhD, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bohr Y, Litwin L, Hankey JR, McCague H, Singoorie C, Lucassen MFG, Shepherd M, Barnhardt J. Evaluating the Utility of a Psychoeducational Serious Game (SPARX) in Protecting Inuit Youth From Depression: Pilot Randomized Controlled Trial. JMIR Serious Games. 2023 Mar 9;11:e38493. doi: 10.2196/38493. PMID 36892940